CLINICAL TRIAL: NCT00105534
Title: A Study to Evaluate the Clinical and Microbial Efficacy and Safety of 1.0 % AzaSite Compared to Vehicle in the Treatment of Bacterial Conjunctivitis
Brief Title: Evaluation of Clinical and Microbial Efficacy and Safety of AzaSite Compared to Vehicle for Bacterial Conjunctivitis (C-01-401-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08635; C-01-401-003
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Bacterial Conjunctivitis
Keywords: Bacterial Conjunctivitis; Pink Eye; Conjunctivitis; Eye Infection; Eye Discharge
MeSH Terms: conditions — Conjunctivitis, Bacterial; Conjunctivitis; Eye Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AzaSite (Experimental)
  Interventions: Drug: AzaSite
- Vehicle (Sham Comparator)
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: AzaSite — 1.0% AzaSite contains 1.0% azithromycin, sodium hydroxide, mannitol, poloxamer 407, citric acid anhydrous, sodium citrate, DuraSite® (polycarbophil, sodium chloride, EDTA disodium and water for injection) and benzalkonium chloride 0.003%. AzaSite was prescribed as a single topical drop to the infected
  eye(s) for 5 days, twice on the first two days (once in the morning and at bedtime) and once a day in the morning (between 7-10 AM) for the following three days.
  Arms: AzaSite
Other: Vehicle — Vehicle contains sodium hydroxide, mannitol, poloxamer 407, citric acid anhydrous, sodium citrate, DuraSite® (polycarbophil, sodium chloride, EDTA disodium and water for injection) and benzalkonium chloride 0.003%. Vehicle was prescribed as a single topical drop to the infected eye(s) for 5 days, twice on the first two days (once in the morning and at bedtime) and once a day in the morning (between 7-10 AM) for the following three days.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the clinical and microbial efficacy and safety of AzaSite compared to vehicle for bacterial conjunctivitis. Adults and children one year of age and older with bacterial conjunctivitis in at least one eye may be eligible. Subjects will be randomly assigned to receive either 1.0 % AzaSite or Vehicle. Three visits will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, of any race, who is at least 1 year of age.
* Subjects must have a clinical diagnosis of acute bacterial conjunctivitis and exhibit mucopurulent or purulent conjunctival discharge (crusty or sticky eyelids, globular and yellow discharge) and redness in at least one eye.
* The symptoms of bacterial conjunctivitis must be present for 3 days (approximately 72 hours) or less.
* Must be willing to discontinue contact lens wear for the duration of the study.

Exclusion Criteria:

* Any uncontrolled, systemic, debilitating disease.
* Use of topical ophthalmic solutions including tear substitutes within 2 hours before and during the study.
* Use of any topical ophthalmic anti-inflammatory agents within 48 hours before and during the study.
* Any active upper respiratory tract infection.
* Pregnant or nursing females.
* Use of any antibiotic (topical or systemic) within 72 hours of enrollment

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2004-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - I Care! Eye Care!, Flagstaff, Arizona
  - Rx For Life, Inc., Cudahy, California
  - North Bay Eye Associates, Petaluma and Santa Rosa, California
  - San Diego Eye and Laser Center, San Diego, California
  - Western States Clinical Research, Wheat Ridge, Colorado
  - Opticare Eye Health Center, Waterbury, Connecticut
  - International Eye Center, Tampa, Florida
  - Welborn Clinic and Welborn Clinic East, Evansville, Indiana
  - Taustine Eye Center, Louisville, Kentucky
  - Bossier Optical Inc., Bossier City, Louisiana
  - Bohn and Joseph Eye Center, Lafayette, Louisiana
  - The Louisiana Eye Center, Zachary, Louisiana
  - Mississippi Eye Associates, Ocean Springs, Mississippi
  - Clinical Research Laboratories, Piscataway, New Jersey
  - Advanced Eyecare and Laser Center, Runnemede, New Jersey
  - Precision Eye Care, Huntington, New York
  - Charlotte Eye, Ear, Nose, and Throat, Charlotte, North Carolina
  - Horizon Eye Center, Charlotte, North Carolina
  - Groat Eyecare Associates, Greensboro, North Carolina
  - Abrams Eye Center, Cleveland, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - University Eye Surgeons, Maryville, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Eye Associates, Nashville, Tennessee
  - Metaclin Research, Inc., Austin, Texas
  - Physicians Eye Associates & Cosmetic Laser, Houston, Texas
  - Marc Sanders, MD, Houston, Texas
  - Mark Mayo, MD, Pasadena, Texas
  - Sun Research Institute, San Antonio, Texas
  - Mountain View Eye Center, Layton, Utah
  - Cottonwood Eye and Laser Clinic, Salt Lake City, Utah
  - Advanced Healthcare, SC, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Abelson MB, Heller W, Shapiro AM, Si E, Hsu P, Bowman LM; AzaSite Clinical Study Group. Clinical cure of bacterial conjunctivitis with azithromycin 1%: vehicle-controlled, double-masked clinical trial. Am J Ophthalmol. 2008 Jun;145(6):959-65. doi: 10.1016/j.ajo.2008.01.019. Epub 2008 Mar 28. PMID 18374301
- See also: Related Info — http://www.insitevision.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AzaSite | Vehicle
Started | 335 | 350
Completed | 313 | 317
Not Completed | 22 | 33
Not completed — Adverse Event | 2 | 5
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 5 | 1
Not completed — Lack of Efficacy | 7 | 15
Not completed — Treatment unmasked | 1 | 0
Not completed — Other Reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- AzaSite; Vehicle: Per protocol population defined as all randomized participants who had administered at least one drop of study drug, who had eye cultures indicating pathogenic bacteria levels as well as the clinical signs of conjunctivitis at Visit 1 and had at least one post first dose clinical assessment.
- Total: Total of all reporting groups
Arm/Group | AzaSite | Vehicle | Total
Number analyzed (Participants) | 130 | 149 | 279
Age Continuous [Mean (Standard Deviation); unit: years] | 25.6 (24.49) | 30.8 (28.07) | 28.4 (26.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 78 | 160
  Male | 48 | 71 | 119

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved Clinical Resolution
Description: Clinical Resolution is defined as absence of all three clinical signs: ocular discharge, bulbar conjunctival injection, and palpebral conjunctival injection.
Time Frame: Visit 3 (Days 6-7)
Population: Per protocol population (defined as all randomized participants who had administered at least one drop of study drug, who had eye cultures indicating pathogenic bacteria levels as well as the clinical signs of conjunctivitis at Visit 1 and had at least one post first dose clinical assessment) with last observation carried forward.
Measure: Number; unit: Participants
Arm/Group | AzaSite | Vehicle
Number analyzed (Participants) | 130 | 149
Participants | 82 | 74

2. Secondary Outcome: Participants Who Achieved Bacteriological Eradication
Description: Bacterial eradication is defined as the eradication of the causative pathogens as indicated by the absence of growth (0 colony forming units/mL) of the original infecting organism(s).
Time Frame: Visit 3 (Day 6-7)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | AzaSite | Vehicle
Number analyzed (Participants) | 130 | 149
Participants | 115 | 99

ADVERSE EVENTS:
Arm/Group | AzaSite | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/333 | 2/350
Other Adverse Events (participants affected / at risk) | 0/333 | 0/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AzaSite (N=333) | Vehicle (N=350)
Cornela Ulcer (Eye disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish, present or use any data or results arising out of the performance of this study for their own instruction, research or publication without the prior express written consent of Sponsor.